CLINICAL TRIAL: NCT03774329
Title: Impact of a Physical Activity Program on Bone Mineral Density (BMD) in Children / Adolescents With Chronic Inflammatory Bowel Disease (IBD): Crohn's Disease, Ulcerative Colitis, Unclassified Chronic Colitis
Brief Title: Impact of a Physical Activity Program on Bone Mineral Density in Children and Adolescents With Chronic Inflammatory Bowel Disease
Acronym: PROPHYSICOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017_04; 2018-A00423-52 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-12-03; First posted 2018-12-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2021-12

CONDITIONS: Crohn's Enteritis; Crohn Disease; Ulcerative Colitis; Chronic; Colitis (Noninfective)
Keywords: inflammatory bowel disease; physical activity; bone mineral density; pediatric
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Bronchiolitis Obliterans Syndrome; Colitis; Inflammatory Bowel Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical activity program (Experimental): Child with an adapted physical activity program
  Interventions: Other: adapted physical activity
- Usual care (Other)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Usual care — Patients included in the control group will not benefit from the intervention in adapted physical activity. However, this will not affect their support. Patients will be seen by their specialist doctor as part of the usual management of their IBD.
  Arms: Usual care
Other: adapted physical activity — Patients in the experimental group will have, in addition to their usual follow-up with their specialist doctor, an intervention in adapted physical activity at home, at the rate of 3 sessions (of a duration of 10 to 20 minutes) per week during 9 consecutive months.
  Arms: physical activity program

SUMMARY:
Muscle and physical activity play an important role in in growth, development and bone health in healthy children, especially during puberty. Children with inflammatory bowel disease (IBD) have lower level and intensity of physical compared to a control group. Several studies have shown that children with IBD have a lower bone mineral density (BMD) than general population, due to risk factors such as corticosteroid use, disease intensity, inflammation, malnutrition and a vitamin D deficiency. This low BMD is associated with an increased risk of fracture. A recent observational study found a positive and significant correlation between BMD in IBD patients and time spent in moderate to vigorous physical activity for one week (unpublished data).The present study aims to show a benefit of an adapted physical activity program on BMD in children and adolescents with IBD.

ELIGIBILITY:
Inclusion Criteria:

* Patient with IBD (Crohn's disease, ulcerative colitis or unclassified chronic colitis) since at least 6 months.
* Computer and internet access at home.
* Consent to adhere to a physical activity program.
* Assent of the child to participation in the research protocol.
* Informed consent of parents or legal guardian.
* Patient benefiting from national health.

Exclusion Criteria:

* At time of inclusion, acute intercurrent events which may lead to a decrease in physical activity (according to the judgment of the investigator) as fractures, recent arthritis, ano-perineal lesions, severe dermatological lesions.
* Chronic, acute or intermittent diseases (other than IBD) that may lead to a decrease in physical activity.
* Refusal of the child to participate to the protocol.
* Refusal of one of the child's parents to participate in the protocol.
* Predictable lack of compliance to study procedures (especially to the physical activity program).
* Child with visual impairment.
* Participation in another interventional study.
* Pregnant or lactating women.
* Patient under protection of justice.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Change in total (whole body) Bone Mineral Density | At 9 months

SECONDARY OUTCOMES:
Change in vertebral BMD | At 9 months
Change in femoral body BMD | At 9 months
Change in time spent (minutes / day) in moderate to vigorous physical activity measured by accelerometry for 7 days | At 9 months
Change in in fat mass measured by two-photon absorptiometry (%) | At 9 months
Change in lean mass measured by two-photon absorptiometry (kg) | At 9 months
Change IMPACT score III | At 9 months
  related quality of life instrument in children with inflammatory bowel disease.
Change in pediatrics crohn's disease activity index or pediatric ulcerative colitis activity index | At 9 months
Change in biologic inflammatory parameters by decrease or increase C-reactive protein | At 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie COOPMAN, MD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - Chu Amiens Picardie, Amiens
  - Hop Jeanne de Flandre Chu Lille, Lille

REFERENCES:
- [Result] Vanhelst J, Coopman S, Labreuche J, Dupont C, Bertrand V, Djeddi D, Turck D, Ley D. Protocol of a randomised controlled trial assessing the impact of physical activity on bone health in children with inflammatory bowel disease. BMJ Open. 2020 May 18;10(5):e036400. doi: 10.1136/bmjopen-2019-036400. PMID 32430452